CLINICAL TRIAL: NCT00910247
Title: Long Term Eslicarbazepine Acetate Extension Study
Brief Title: Eslicarbazepine Acetate Monotherapy Long Term Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 093-050
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Epilepsy
Keywords: Seizures; Epilepsy; Anticonvulsant; Monotherapy; Epilepsy with simple or complete partial onset seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — eslicarbazepine acetate

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- eslicarbazepine acetate (Experimental): Open-label treatment with eslicarbazepine acetate will be at doses between 800 and 2400 mg QD
  Interventions: Drug: Eslicarbazepine acetate

INTERVENTIONS:
Drug: Eslicarbazepine acetate — 800 to 2400 mg once daily (QD)
  Other Names: SEP-0002093; BIA 2-093

SUMMARY:
This is a long term, open-label, safety extension study in subjects with partial onset seizures.

DETAILED DESCRIPTION:
This is a long term, multicenter, open-label, safety extension study in subjects with partial onset seizures who have just completed, discontinued, or exited the 18-week treatment phase of Protocols 093-045 or 093-046. The initial study duration is 1 year with the option of continuing study drug treatment post 1 year until a subject discontinues study, the study drug becomes clinically available in the subject's locale, or the sponsor terminates the study drug clinical development program.

This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Subject Inclusion/Exclusion Criteria:

* Subject who completed, exited, or discontinued for reasons other than safety from the 18-week treatment phase of Protocols 093-045 or 093-046 and are willing to continue participation in this study are eligible. Subject must have completed at least the first 3 weeks of the 18-week double-blind treatment period of Protocols 093-045 or 093-046 to be eligible.
* Subject must give written informed consent prior to participation in the study. For subjects <18 years of age, the informed consent must be signed by the subject's parent or legal guardian, and, when appropriate and/or required by state or local law, minor subjects must give written informed assent prior to participation in the study. All subjects must sign privacy authorization form, if applicable. All females of child bearing potential (≤65 years of age) must also sign the "Women of Childbearing Potential" Addendum.
* Subjects must, in the opinion of the Investigator (with consultation with Medical Monitor as appropriate), continue to potentially benefit from continued study participation and have no new medical conditions that would preclude study participation.
* If female subject, must continue the accepted method of birth control defined in Protocols 093-045 or 093-046 for the duration of this study as well
* Criterion for Continuation into the Post 1 year Part of Study:

For subjects to continue into the post 1 year part of the study, subjects must, in the opinion of the Investigator (with consultation with Medical Monitor, as appropriate), continue to potentially benefit from continued study participation and have no new medical conditions that would preclude study participation.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2009-08; Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sunovion Pharmaceuticals
Locations (122):
- United States (96):
  - Neurology Clinic, P.C., Northport, Alabama
  - 21st Century Neurology, a division of Xenoscience, Inc., Phoenix, Arizona
  - Clinical Research Consortium-Arizona, Phoenix, Arizona
  - Arizona Neurological Institute, Sun City, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - University of Arizona, Health Sciences Center, Tucson, Arizona
  - Arkansas Neurology, Conway, Arkansas
  - K&S Professional Research Services, LLC, Little Rock, Arkansas
  - Sutter East Bay Medical Foundation, Berkeley, California
  - Neuro-Pain Medical Center, Fresno, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - Faculty of Physicians and Surgeons of Loma Linda University, Loma Linda, California
  - Viking Clinical Research Center, Murrieta, California
  - Viking Clinical Research, Murrieta, California
  - Northridge Neurological Research Center, Northridge, California
  - Yafa Minazad, Pasadena, California
  - Neurological Research Institute, Santa Monica, California
  - Collaborative Neuroscience Network, Torrance, California
  - Neurosearch II Inc, Ventura, California
  - Neurosciences Clinic - University of Colorado Hospital, Aurora, Colorado
  - Denver Health, Denver, Colorado
  - Associated Nuerologists, PC, Danbury, Connecticut
  - JEM Research, LLC, Atlantis, Florida
  - Bradenton Clinical Research, Bradenton, Florida
  - Miami Research Inc., Coral Gables, Florida
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Neurology Associates, Maitland, Florida
  - San Marcus Research Clinic, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Neuroscience Consultants, Miami, Florida
  - Pediatric Neurology, PA, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Bay Neurological Institute, Panama City, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Pediatric Epilepsy & Neurology Specialists, PA, Tampa, Florida
  - Palm Beach Clinical Research Network, LLC, Wellington, Florida
  - PANDA Neurology and Atlanta Heachache Specialists, Atlanta, Georgia
  - Harbin Clinic, Rome, Georgia
  - Consultants in Epilepsy and Nuerology, Boise, Idaho
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - J.W.M. Neurology P.C., Indianapolis, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Bluegrass Epilepsy Research, LLC, Lexington, Kentucky
  - ECommunity Research LLC, Hammond, Louisiana
  - MMP Neuroloy, Scarborough, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Wayne State University/Detroit Medical Center, Detroit, Michigan
  - Minneappolis Clinic of Neurology, Golden Valley, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - University Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - UMDNJ DOC 8th Floor 8100, Newark, New Jersey
  - Five Towns Neuroscience Research, Cedarhurst, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Department of Neurology, Winston-Salem, North Carolina
  - Ohio Clinical Research Partners, LLC, Canton, Ohio
  - The University of Toledo Health Science Campus, Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Tulsa Clinical Research LLC, Tulsa, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Dept of Neurology, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Gus Stratton / Neurology, Cranston, Rhode Island
  - VU Department of Neurology, Nashville, Tennessee
  - Neurology Associates of Arlington, P.A., Arlington, Texas
  - Edwin A Green, Jr., MD, Brownwood, Texas
  - Texas Neurology, PA, Dallas, Texas
  - Neurological Clinic of Texas, P.A., Dallas, Texas
  - UT Health Science Center at Houston/ Dept of Neurology, Houston, Texas
  - MD, Houston, Texas
  - Neurology Associates of Arlington, P.A., Mansfield, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Road Runner Research, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Utah Department of Neurology, Salt Lake City, Utah
  - Neurological Associates of Washington, Bellevue, Washington
  - Rainier Clinical Research Center Inc., Renton, Washington
  - Pacific Medical Centers, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Regional Epilepsy Center, Milwaukee, Wisconsin
- Bulgaria (4):
  - Multiprofile Hospital for Active Treatment "Pulse," AD, Town of Blagoegrad, Blagoevgrad
  - Univesity Multiprofile Hospital for Active Treatment "Dr. George Stranski," EAD, town of Pleven, Pleven
  - Second Multiprofile Hospital for Active Treatment, Sofia
  - Diagnostic and Consultative Center "Equita" EOOD, town of Varna Neurology office, Varna
- Canada (3):
  - London Health Sciences Centre, University Campus, London, Ontario
  - Neuro-Epilepsy Clinic/ Neuro Rive-Sud, Greenfield Park, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Czechia (6):
  - Policlinic Chocen, Private Neurology, Smetanova Lhota, Chocen
  - Cerebrovaskularni poradna s.r.o, Třebovice, Ostrava
  - CTC Rychnov nad Kneznou, Rychnov nad Kněžnou, Praugue
  - Evzen Nespor, Prague, Strasnice
  - Poradna pro epilepsie, Koty, Zlín
  - Neurologicka ordinance, Prague
- Serbia (2):
  - Clinic of Neurology, Clinical Center of Serbia, Belgrade
  - Institute of Mental Health, Department of epilepsy and clinical neurophysiology, Belgrade
- Ukraine (11):
  - Communal Institution "Dnipropetrovsk Regional Clinical Hospital named after l.l. Mechnikov" Regional Center of psychosomatic disorders, Psychoneurology department for patients with psychosomatic disorders and borderline conditions, Dnipropetrovsk
  - Communal Medical and Preventive Treatment Institution "Regional Clinical Psychiatric Hospital" Donetsk National Medical University, Donetsk
  - State Treatment and Prevention Institution " Central clinical hospital of Ukrzalizntysya" Neurology Department of Neuropathology and Child Neurology, Kharkiv
  - State Institution "Institute of neurology, psychiatry, and narcology of AMS of Ukraine" Department of cerebrovascular patology, Kharkiv
  - State Institution "Institute of the Health Care of Children and Adolescents of Academy of Medical Sciences of Ukraine Dept of Psych, Kharkiv
  - State Institution Railway Clinical Hospital #1 of Kiev Railway Station of DTGO South Western Railroad Psycho-neurological Department, Kiev
  - Communal Institution "Lviv Regional Clinical Psych Hospital", Lviv
  - Communal Institution "Odessa Regional Clinical Psych Hospital #1" Department of Day Care, Odesa
  - Poltava Regional Clinical Psychiatric Hospital named O.F. Maltsev, Poltava
  - Crimean Republican Institution "Clinical Psychiatric Hospital #1", Simferopol
  - Communal Institution "Vinnystsia Regional Psycho-Neurological Hospital named after O.I. Yuschenko, Vinnytsia National Medical University named after M.I. Pirogov, Dispensary department, Department of Psychiatry and Addictology, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects that participated in either study 093-045NCT00866775) or study 093-046(NCT01091662) were eligible to participate in study 093-050
Pre-assignment Details: Subjects who completed the 18-week treatment period or exited the study per protocol may be eligible to participate. Subjects who discontinued for reasons other than reaching the exit criteria may be eligible if there is no safety concern, however, subjects must have completed at least the first 3 weeks of the 18-week double-blind treatment
Period: Overall Study
Arm/Group | Eslicarbazepine Acetate
Started | 274
Completed | 205
Not Completed | 69
Not completed — Adverse Event | 15
Not completed — Death | 2
Not completed — Lost to Follow-up | 10
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 10
Not completed — Withdrawal by Subject | 25
Not completed — Not collected | 4

BASELINE CHARACTERISTICS:
Population: full analysis set
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 258
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134
  Male | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 246
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 229
  More than one race | 2
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  Canada | 3
  United States | 167
  Czechia | 27
  Ukraine | 57
  Bulgaria | 18
  Serbia | 2

OUTCOME MEASURES:

1. Primary Outcome: Number and Percent of Subjects With Treatment Emergent Adverse Events
Description: Number and percent of subjects with treatment emergent adverse events
Time Frame: One year
Population: The Intent-to -Treat (ITT) population consisted of all subjects who had taken any open-label study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
Participants | 220

2. Secondary Outcome: Number and Percentage of Subjects With Potentially Clinically Significant Clinical Laboratory Evaluations
Description: Number and percentage of subjects with potentially clinically significant clinical laboratory evaluations
Time Frame: 1 year
Population: The intent-to-treat (ITT) population consisted of all subjects who have taken any open-label study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
Participants | 186

3. Secondary Outcome: Number and Percent of Subjects With Normal Baseline Sodium Reaching Blood Sodium ≤135 mmol/L, ≤130 mmol/L, and ≤125 mmol/L
Description: Number and percentage of subjects who had normal sodium value (i.e. >135 mEq/L) at baseline but reached <=135 mEq/L and >130 mEq/L, <=130 mEq/L and >125 mEq/L, or <=125 mEq/L at any post baseline.
Time Frame: 1 year
Population: ITT subjects with baseline sodium and at least one post baseline sodium value
Measure: Count of Participants; unit: Participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 261
Participants
  <=135 mEq/L and >130 mEq/L | 48
  <=130 mEq/L and >125 mEq/L | 22
  <=125 mEq/L | 4

4. Secondary Outcome: Percentage of Subjects With Increase of Body Weight ≥7%
Description: Percentage of subjects with increase of body weight ≥7%
Time Frame: 1 year
Population: The intent-to-treat (ITT) population consisted of all subjects who have taken any open-label study medication.
Measure: Number; unit: percentagae of participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
percentagae of participants | 27

5. Secondary Outcome: Number and Percentage of Subjects With Orthostatic Effects.
Description: Number and percentage of subjects with orthostatic effects.
Time Frame: 1 year
Population: The intent-to-treat (ITT) population consisted of all subjects who have taken any open-label study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
Participants | 67

6. Secondary Outcome: Number and Percentage of Subjects With QTc-F Changes (in Categories) From Baseline.
Description: Number and percentage of subjects by QT interval corrected using the Fridericia fomula (QTcF) categories
  Based on the numbers of subjects who had at least one post-baseline assessment, the number and percentage of subjects with QTcF values in the following categories were summarized:
  1. >500 millisecond (msec) at any post-baseline timepoint but not present at baseline
  2. >480 msec at any post-baseline timepoint but not present at baseline
  3. >450 msec at any post-baseline timepoint but not present at baseline
  4. Change from Baseline >=60 ms for at least one post-baseline measurement
  5. Change from Baseline >=30 ms for at least one post-baseline measurement and <60 ms for all post-baseline measurement
  QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle.
Time Frame: Baseline, Month 12
Population: The intent-to-treat (ITT) subjects with at least one post-baseline assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 272
Participants
  >500ms at any postbaseline not present at baseli | 0
  >450ms at any postbaseline not present at baseline | 9
  >480ms at any postbaseline not present at baseline | 1
  CFB >=60 ms for at least one post-baseline | 0
  CFB>=30ms for at least one &<60ms for all PBL | 42

7. Secondary Outcome: Percentage of Events in Each Classification of the Columbia Suicide Severity Rating Scale (C SSRS).
Description: The C-SSRS is an instrument designed to systematically assess and track suicidal behavior and suicidal ideation. The C-SSRS will be completed by the Investigator or Sub-Investigator (or qualified site personnel).
  Suicidal ideation is collected as any occurrence of wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intent to act, active suicidal ideation with some intent to act, without specific plan, active suicidal ideation with specific plan and intent.
  Suicidal behavior is collected as any occurrence of actual attempts, Non-Suicidal Self-Injurious Behavior, interrupted attempts, aborted attempts, or preparatory acts or behavior, suicidal behavior.
  Any suicidality is defined as having at least one occurrence of Suicidal Behavior or Suicidal Ideation.
Time Frame: 1 year
Population: The Intent-to-Treat (ITT) population consisted of all subjects that received any open-label study medication
Measure: Number; unit: percentage of events
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
percentage of events
  Any Suicidality | 4.0
  Any suicidal behavior | 0.7
  Any suicidal ideation | 3.6

8. Secondary Outcome: Time on Eslicarbazepine Acetate Monotherapy.
Description: The start of the monotherapy period was defined as the date of termination of all other anti-epileptic drugs while taking study medication. Time on eslicarbazepine acetate monotherapy is defined from the date of the first monotherapy dose in 093-045 or 093-046 study to the last known dose of monotherapy treatment, regardless of dose change and the time gap between the parent studies and the current study.
Time Frame: One year
Population: ITT Subjects who started the monotherapy period (Visit 6/Week 8) in 093-045 or 093-046 and did not add a non-rescue/emergency Antiepileptic drug (AED) during the start date of the monotherapy period
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 238
Days | NA [NA to NA] — Median not calculable due to lack of events

9. Secondary Outcome: Change in Seizure Frequency From Baseline.
Description: Relative (%) change in standard seizure frequency(SSF) from baseline
Time Frame: Month 12 from baseline
Population: Intent-to-treat (ITT) population consisted of all subjects who had taken any open-label study medication
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
percent change | -66.4 [-88.8 to -32.3]

10. Secondary Outcome: Responder Rate (Percentage of Subjects With a ≥50% Reduction of Seizure Frequency From Baseline).
Description: Responder rate (percentage of subjects with a ≥50% reduction of seizure frequency from baseline).
Time Frame: One year
Population: The intent-to-treat (ITT) population consisted of all subjects who have taken any open-label study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
percentage of participants | 62.4

11. Secondary Outcome: Percentage of Subjects That Are Seizure-free During Study
Description: Percentage of subjects that are seizure-free during study
Time Frame: 1 year
Population: The intent-to-treat (ITT) population consisted of all subjects who have taken any open-label study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
percentage of participants | 7.3

12. Secondary Outcome: Completion Rate (% of Subjects Completing the One Year Treatment)
Description: Completion rate (% of subjects completing the one year treatment)
Time Frame: One year
Population: The intent-to-treat (ITT) population consisted of all subjects who have taken any open-label study medication.
Measure: Number; unit: percentagae of participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
percentagae of participants | 74.8

13. Secondary Outcome: Treatment Retention Time (Time to Withdrawal Due to Lack of Efficacy or Adverse Events)
Description: The retention time is defined from the start of eslicarbazepine acetate monotherapy period in 093-045 or 093-046 to the last known dose of open-label eslicarbazepine acetate. The time may include taking eslicarbazepine acetate concomitantly with other anti-epileptic drugs. If a subject's termination reason(s) includes: withdrawal of consent, lost to follow-up, physician decision or other, then it was assumed the subject terminated the study due to lack of efficacy.
Time Frame: One year
Population: Intent-to-treat (ITT) subjects who started the monotherapy period in 093-045 or 093-046 (visi t6/week 8)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 255
days | NA [NA to NA] — Median time in Days is NA so the 95% CI cannot be calculated since median not calculable due to lack of events during the 1 year open-label period.

14. Secondary Outcome: Change in Total Score From Baseline in 31-Item Quality of Life in Epilepsy (QOLIE-31).
Description: Change in the overall score from baseline in 31-Item Quality of Life in Epilepsy (QOLIE-31 )
  The QOLIE-31 overall score was obtained by using a weighted average of multi-item scale scores. The recorded responses were converted to 0-100 point scales. The mean of the individual item scores in each subgroup were calculated, with higher converted scores reflecting better quality of life.
Time Frame: baseline and Month 12
Population: The intent-to-treat (ITT) population consisted of all subjects who have taken any open-label study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
units on a scale | 6.6 (15.29)

15. Secondary Outcome: Change in Total Score From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS).
Description: The total score of MADRS is defined as the sum of all individual item scores. Each of the 10 symptoms of depression on MADRS is measured on a scale of 0 to 6 with 0 representing the lowest severity of the symptom and 6 representing the highest severity.
Time Frame: 1 year
Population: The intent-to-treat (ITT) population consisted of all subjects who have taken any open-label study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
units on a scale | -1.5 (6.17)

16. Secondary Outcome: Change in Total Score From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) in Those Subjects With a MADRS Score of ≥14 at Screening
Description: The total score of MADRS is defined as the sum of all individual item scores . Each of the 10 symptoms of depression on MADRS is measured on a scale of 0 to 6 with 0 representing the lowest severity of the symptom and 6 representing the highest severity.
Time Frame: baseline and Month 12
Population: The intent-to-treat (ITT) population consisted of all subjects who have taken any open-label study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 274
units on a scale | -1.5 (6.17)

17. Secondary Outcome: Completion Rate (% of Subjects Completing Each Visit Post-one Year).
Description: Completion rate (% of subjects completing each visit post-one year).
Time Frame: post 1 year
Population: The intent-to-treat (ITT) subjects who entered the post - 1- year open -label period.
Measure: Number; unit: percentagae of participants
Arm/Group | Eslicarbazepine Acetate
Number analyzed (Participants) | 198
percentagae of participants | 66.7

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Eslicarbazepine Acetate
All-Cause Mortality (participants affected / at risk) | 2/274
Serious Adverse Events (participants affected / at risk) | 32/274
Other Adverse Events (participants affected / at risk) | 166/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eslicarbazepine Acetate (N=274)
sinus tachycardia (Cardiac disorders) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1)
abdominal pain upper (Gastrointestinal disorders) | 1 (1)
colitis (Gastrointestinal disorders) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
non-cardiac chest pain (General disorders) | 3 (3)
irritability (General disorders) | 1 (1)
sudden unexplained death in epilepsy (General disorders) | 1 (1)
cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1)
chronic sinusitis (Infections and infestations) | 1 (1)
histoplasmosis (Infections and infestations) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
tooth infection (Infections and infestations) | 1 (1)
accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
collapse of lung (Injury, poisoning and procedural complications) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)
post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1)
electroencephalogram (Investigations) | 1 (1)
failure to thrive (Metabolism and nutrition disorders) | 1 (1)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
non-small cel lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
partial seizures with secondary generalisation (Nervous system disorders) | 7 (7)
complex partial seizures (Nervous system disorders) | 3 (3)
simple partial seizures (Nervous system disorders) | 2 (2)
akathisia (Nervous system disorders) | 1 (1)
grand mal convulsion (Nervous system disorders) | 1 (1)
postictal paralysis (Nervous system disorders) | 1 (1)
status epilepticus (Nervous system disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
suicidal ideation (Psychiatric disorders) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 1 (1)
emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
accelerated hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eslicarbazepine Acetate (N=274)
nausea (Gastrointestinal disorders) | 24 (31)
vomiting (Gastrointestinal disorders) | 16 (20)
diarrhoea (Gastrointestinal disorders) | 15 (19)
fatigue (General disorders) | 23 (25)
nasopharyngitis (Infections and infestations) | 24 (35)
influenza (Infections and infestations) | 14 (15)
fall (Injury, poisoning and procedural complications) | 20 (33)
back pain (Musculoskeletal and connective tissue disorders) | 16 (16)
headache (Nervous system disorders) | 64 (144)
dizziness (Nervous system disorders) | 46 (81)
complex partial seizures (Nervous system disorders) | 14 (18)
depression (Psychiatric disorders) | 18 (19)
insomnia (Psychiatric disorders) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT00910247/SAP_000.pdf
  • Study Protocol: Final (2013-06-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT00910247/Prot_001.pdf
  • Study Protocol: Amendment history (2013-11-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT00910247/Prot_002.pdf